CLINICAL TRIAL: NCT02221167
Title: Rx Milk: Donor Milk Supplementation to Increase Breastfeeding Duration & Exclusivity, a Randomized Controlled Trial
Brief Title: Rx Milk Study of Donor Milk Supplementation to Improve Breastfeeding Outcomes
Acronym: Rx Milk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laura Kair (Other)
Collaborators: Children's Miracle Network (Other); The Gerber Foundation (Other)
Responsible Party: Sponsor-Investigator, Laura Kair, Adjunct Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 201406730
Record Dates: First submitted 2014-08-18; First posted 2014-08-20 (Estimated); Last update posted 2018-03-16 (Actual); Status verified 2018-03

CONDITIONS: Breastfeeding Duration; Exclusive Breastfeeding; Donor Milk Supplementation
Keywords: breastfeeding; donor milk; formula; exclusive breastfeeding; newborn
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exclusive breastfeeding (No Intervention): Infants in the exclusive breastfeeding group will continue to breastfeed.
- Donor Milk (Active Comparator): Infants in this arm will continue to breastfeed and will be given 10 ml of donor breast milk by syringe after each breastfeeding until their mother's milk "comes in." (until the onset of lactogenesis II)
  Interventions: Other: Donor Milk

INTERVENTIONS:
Other: Donor Milk — breastfeeding plus 10 ml of donor milk by syringe after each breastfeeding until mother's milk "comes in."
  Other Names: donor breast milk; human donor milk
  Arms: Donor Milk

SUMMARY:
This study is a randomized controlled trial seeking to determine whether supplementing infants at risk for excessive neonatal weight loss with a small volume of human donor milk prophylactically in the first 1-3 days of life, before maternal mature milk production (before mom's milk "comes in") will decrease the incidence of formula use at 1 week and 1, 2, and 3 months of life and increase the rate of exclusive breastfeeding in this high-risk population.

We hypothesize that supplementation of term infants who have lost greater than or equal to 5% birth weight by 36 hours of age with a small volume of donor breast milk following feeds, until mature milk production, will result in decreased supplemental formula use at 1 week and increased exclusive as well as any breastfeeding at 1 week and 1, 2, and 3 months. This study's specific aims are to compare the effectiveness of encouraging in-hospital exclusive breastfeeding with offering early small-volume donor milk supplementation in a population of infants at risk for excessive neonatal weight loss with goals of 1) decreasing the incidence of formula supplementation at 1 week of life and 2) improving breastfeeding duration.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age greater than or equal to 37 weeks
* Weight loss greater than or equal to 5% (rounded to nearest whole percent) of birth weight in the first 36 hours after birth
* Chronologic age of 24-48 hours old at the time of study enrollment

Exclusion Criteria:

* twins and higher level multiples
* infant has congenital or chromosomal anomalies that may affect feeding, diagnosed prior to study enrollment
* mother incarcerated
* mother's age <18 years
* mother reports mature milk production prior to study enrollment
* mother does not speak English
* infants offered > 1 supplemental feeding of formula or donor milk
* weight loss greater than 10%

Ages: 24 Hours to 48 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2014-07; Primary Completion 2016-07 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Any formula use at 1 week of age | 1 week
  Any formula intake within the last 24 hours.

SECONDARY OUTCOMES:
Exclusive breastfeeding | 3 months
  Infants receiving breast milk and no formula in the last 24 hours.
Any breastfeeding at 3 months | 3 months
  Infants receiving some breast milk in addition to some formula in the last 24 hours.
Any breastfeeding | 1 month
Exclusive breastfeeding | 1 month
Exclusive breastfeeding | 2 months
Any breastfeeding | 2 months
Any breastfeeding | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Laura R Kair, MD, Principal Investigator — University of Iowa; Tarah T Colaizy, MD, MPH, Study Director — University of Iowa; Valerie J Flaherman, MD, MPH, Study Director — University of California, San Francisco
Locations (1):
- University of Iowa Children's Hospital, Iowa City, Iowa, United States

REFERENCES:
- [Background] Flaherman VJ, Aby J, Burgos AE, Lee KA, Cabana MD, Newman TB. Effect of early limited formula on duration and exclusivity of breastfeeding in at-risk infants: an RCT. Pediatrics. 2013 Jun;131(6):1059-65. doi: 10.1542/peds.2012-2809. Epub 2013 May 13. PMID 23669513
- [Background] Flaherman VJ, Kuzniewicz MW, Li S, Walsh E, McCulloch CE, Newman TB. First-day weight loss predicts eventual weight nadir for breastfeeding newborns. Arch Dis Child Fetal Neonatal Ed. 2013 Nov;98(6):F488-92. doi: 10.1136/archdischild-2012-303076. Epub 2013 Jul 17. PMID 23864443
- [Background] Flaherman VJ, Bokser S, Newman TB. First-day newborn weight loss predicts in-hospital weight nadir for breastfeeding infants. Breastfeed Med. 2010 Aug;5(4):165-8. doi: 10.1089/bfm.2009.0047. PMID 20113202
- [Derived] Kair LR, Flaherman VJ, Colaizy TT. Effect of Donor Milk Supplementation on Breastfeeding Outcomes in Term Newborns: A Randomized Controlled Trial. Clin Pediatr (Phila). 2019 May;58(5):534-540. doi: 10.1177/0009922819826105. Epub 2019 Jan 28. PMID 30688082
- See also: Baby Friendly USA — http://www.babyfriendlyusa.org/about-us/baby-friendly-hospital-initiative/the-ten-steps